CLINICAL TRIAL: NCT03448198
Title: Validation of a New Technique for the Evaluation of the Patello-femoral Joint Kinematics
Acronym: CINE-FEMORO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Claudio Belvedere, PhD, Istituto Ortopedico Rizzoli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 39521/2012
Record Dates: First submitted 2018-02-09; First posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Knee Osteoarthritis
Keywords: total knee arthroplasty; patellar resurfacing; patellar tracking; patello-femoral joint kinematics; surgical navigation; computer-aided surgery
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Masking Description: open label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Knee arthritis (Other): Total knee replacement
  Interventions: Procedure: Total knee replacement

INTERVENTIONS:
Procedure: Total knee replacement — Primary knee gonarthrosis treated with navigated total knee replacement and computer-assisted patellar replacement.

SUMMARY:
The objective of this study is to validate a new technique for intraoperative quantification of the patello-femoral joint kinematics in patients undergoing total knee replacement, and for postoperative quantification of implanted knee and general lower limb activity, along with relevant muscle dynamics.

DETAILED DESCRIPTION:
In total knee replacement with patellar resurfacing, the patellar bone preparation and relevant component positioning, including relevant motion assessments, are still not navigated, and only femoral/tibial component positioning is supported by computer-assistance. After surgery, anterior knee pain is generally reported and this may due to prosthesis component mal-positioning, including the patella, and, ultimately, this may result in revision arthroplasty. Within computer-assisted surgery, surgical navigated system have been introduced to monitor femur and tibia prosthesis implantation and to assess tibio-femoral joint kinematics. In this context, the patella is still disregarded or limitedly considered, whereas it is still debated if the patella should be resurfaced in total knee replacement. Recently, new navigation-based procedures have been tested to allow the intra-operative monitoring of patellar-based data for more proper patellar resurfacing; at follow-up under active conditions, video-fluoroscopy, so far used to assess general tibio-femoral kinematics, offers the potentials for patellar motion tracking.

The possibility in vivo to perform intra-operative evaluations of the patello-femoral joint data, i.e. including patellar bone morphology and motion, via computer assisted procedures during surgery would allow the surgeon to have a more complete comprehension of the knee functioning in patients undergoing total knee replacement; these procedures, along with derived data, can act as a support in for the most critical surgical actions in terms of femoral/tibial prosthesis component implantation and related patellar resurfacing. Furthermore, at post-operative follow-ups via fluoroscopic acquisitions and gait analysis, it is possible to evaluate how the implant is able to recover, or not, the normative physiological motion at both tibio-femoral and patello-femoral joint.

The goal of this study is to validate a new technique for intra-operative quantification of the patello-femoral joint kinematics in patients undergoing total knee replacement, and for postoperative quantification of implanted knee and general lower limb activity, along with relevant muscle dynamics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral primary knee arthrosis indicated for total knee replacement.
* Patients able to understand the protocol and to sign the informed consent.

Exclusion Criteria:

* Patients with indications for revision surgery.
* Patients with patellectomy.
* Child-bearing female.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-11-16 (Actual); Primary Completion 2014-05-16 (Actual); Study Completion 2014-11-16 (Actual)

PRIMARY OUTCOMES:
Knee prosthesis rotational alignment | At time of surgery
  Rotational (in deg) positioning of femur, tibia and patella prosthesis components.
Knee prosthesis translational alignment | At time of surgery
  Translational (in mm) positioning of femur, tibia and patella prosthesis components.

SECONDARY OUTCOMES:
Intra-operative knee joint rotations | At time of surgery
  Assessed rotations (in deg): tibio-femoral flexion-extension, ad-abduction and internal-external rotation; patello-femoral flexion-extension, medio-lateral rotation and tilt.
Intra-operative knee joint translations | At time of surgery
  Assessed translations (in mm): tibio-femoral and patello-femoral anterio-posterior, medial-lateral and proximal-distal translations.
Post-operative knee joint rotations | 24 months
  Assessed rotations (in deg): tibio-femoral flexion-extension, ad-abduction and internal-external rotation; patello-femoral flexion-extension, medio-lateral rotation and tilt.
Post-operative knee joint translations | 24 months
  Assessed translations (in mm): tibio-femoral and patello-femoral anterio-posterior, medial-lateral and proximal-distal translations.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ensini, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Cutbill JW, Ladly KO, Bray RC, Thorne P, Verhoef M. Anterior knee pain: a review. Clin J Sport Med. 1997 Jan;7(1):40-5. doi: 10.1097/00042752-199701000-00008. PMID 9117525
- [Background] Sparmann M, Wolke B, Czupalla H, Banzer D, Zink A. Positioning of total knee arthroplasty with and without navigation support. A prospective, randomised study. J Bone Joint Surg Br. 2003 Aug;85(6):830-5. PMID 12931800
- [Background] Belvedere C, Catani F, Ensini A, Moctezuma de la Barrera JL, Leardini A. Patellar tracking during total knee arthroplasty: an in vitro feasibility study. Knee Surg Sports Traumatol Arthrosc. 2007 Aug;15(8):985-93. doi: 10.1007/s00167-007-0320-1. Epub 2007 Apr 13. PMID 17431587
- [Background] Burnett RS, Haydon CM, Rorabeck CH, Bourne RB. Patella resurfacing versus nonresurfacing in total knee arthroplasty: results of a randomized controlled clinical trial at a minimum of 10 years' followup. Clin Orthop Relat Res. 2004 Nov;(428):12-25. PMID 15534514
- [Background] Fantozzi S, Benedetti MG, Leardini A, Banks SA, Cappello A, Assirelli D, Catani F. Fluoroscopic and gait analysis of the functional performance in stair ascent of two total knee replacement designs. Gait Posture. 2003 Jun;17(3):225-34. doi: 10.1016/s0966-6362(02)00096-6. PMID 12770636

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2012-11-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT03448198/Prot_SAP_ICF_000.pdf